CLINICAL TRIAL: NCT00002643
Title: INTENSIVE THERAPY WITH GROWTH FACTOR SUPPORT FOR PATIENTS WITH EWING'S TUMOR METASTATIC AT DIAGNOSIS: A PEDIATRIC ONCOLOGY GROUP PHASE II STUDY
Brief Title: Combination Chemotherapy in Treating Patients With Newly Diagnosed Metastatic Ewing's Sarcoma or Primitive Neuroectodermal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01832; POG-9457; CCG-P9457; CDR0000064137 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-06-18 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2007-03

CONDITIONS: Neutropenia; Sarcoma
Keywords: neutropenia; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Neutropenia; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Filgrastim; Amifostine; Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Topotecan; Vincristine

ARMS (1):
- Arm I (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: topotecan hydrochloride; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: topotecan hydrochloride
Drug: vincristine sulfate
Procedure: conventional surgery
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
Phase II trial to study the effectiveness of combination chemotherapy in treating patients with newly diagnosed metastatic Ewing's sarcoma or primitive neuroectodermal tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the response rate and duration of response of patients with newly diagnosed, metastatic Ewing's sarcoma or primitive neuroectodermal tumor treated with maximally intensified VAdrC (vincristine, doxorubicin, cyclophosphamide) alternating with IE (ifosfamide, etoposide).

II. Evaluate the response to new agents (first topotecan, then topotecan with cyclophosphamide) utilized in an upfront treatment window.

III. Assess the role of surgery with regard to local control of primary and metastatic sites and disease course.

IV. Evaluate whether individual variability in ifosfamide and cyclophosphamide metabolism correlates with toxicity and/or response.

V. Evaluate the rise in the absolute neutrophil count following one dose of filgrastim (G-CSF) given immediately prior to a chemotherapy course as an indicator of bone marrow reserve and subsequent myelosuppression.

VI. Determine if amifostine provides significant chemo-radio protection, particularly against the cumulative toxicities of this intensive therapy.

OUTLINE: This is a partially randomized, multicenter study.

Patients are treated on the investigational window first or proceed to induction therapy immediately, if aggressive treatment is necessary.

INVESTIGATIONAL WINDOW: Patients receive cyclophosphamide IV and topotecan IV over 30 minutes on days 1-5. Filgrastim (G-CSF) is administered subcutaneously (SQ) beginning day 6 until blood cell counts recover. Treatment is repeated at week 3.

INDUCTION THERAPY: Patients over 12 months old are randomized to receive amifostine or not. Patients receive etoposide IV over 45 minutes and ifosfamide IV over 2 hours on days 1-5. Amifostine IV over 15 minutes is also administered prior to ifosfamide. Patients receive G-CSF SQ (or IV over 2 hours) beginning on day 6. This course of treatment is administered on weeks 6, 12, and 18. Patients receive the VAdrC chemotherapy regimen on weeks 9 and 15. This regimen consists of vincristine IV and amifostine IV over 15 minutes on days 1, 8, and 15, cyclophosphamide IV over 30 minutes and doxorubicin IV over 48 hours on days 1 and 2, and G-CSF beginning on day 3. The VAdrC regimen is continued during local therapy on weeks 21-29 and 39-47, except the day 15 dose of vincristine is omitted, cyclophosphamide is administered on day 1 only on weeks 21, 24, 27, 39, 42, and 45, and doxorubicin is replaced with etoposide IV over 60 minutes on days 1-3 on weeks 24, 28, 42, and 45. Local therapy begins after 21 weeks of chemotherapy. Patients who respond to chemotherapy and have resectable disease undergo a complete resection with negative margins. Patients with unresectable disease or bulky lesions undergo radiotherapy. Some patients may undergo both surgery and radiotherapy. Local therapy of metastases is delayed until after week 39. Patients are followed every 3 months for 1 year, every 6 months for 2 years, then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed, pathologically confirmed Ewing's sarcoma or primitive neuroectodermal tumor (PNET)
* Diagnosis established from biopsy of primary tumor Light microscopy (hematoxylin and eosin stained) consistent with Ewing's sarcoma or PNET
* No immunohistochemical or ultrastructural characteristics inconsistent with Ewing's sarcoma or PNET or suggestive of rhabdomyosarcoma
* Metastatic disease required
* Biopsy of radiographically questionable metastases (e.g., pulmonary lesions) required
* Chest wall tumor with separate pleural mass considered metastatic
* No positive pleural fluid cytology alone

PATIENT CHARACTERISTICS:

* Age: 30 and under
* Absolute neutrophil count greater than 1,200/mm3
* Platelet count greater than 120,000/mm3
* Bilirubin less than 1.5 mg/dL
* AST/ALT less than 3 times normal
* Creatinine normal for age
* Significant renal abnormality/disease eligible only if nuclear GFR is normal and study coordinator approves
* Echocardiogram or MUGA normal

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* Resection at diagnosis is discouraged but does not exclude

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 1995-04; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark L. Bernstein, MD, FRCPC, Study Chair — Montreal Children's Hospital at McGill University Health Center; Paul A. Meyers, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (49):
- United States (43):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Via Christi Regional Medical Center-Saint Francis Campus, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Mission Hospital, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia
  - Montreal Children's Hospital, Montreal, Quebec
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland

REFERENCES:
- [Background] Souid AK, Fahey RC, Dubowy RL, Newton GL, Bernstein ML. WR-2721 (amifostine) infusion in patients with Ewing's sarcoma receiving ifosfamide and cyclophosphamide with mesna: drug and thiol levels in plasma and blood cells, a Pediatric Oncology Group study. Cancer Chemother Pharmacol. 1999;44(6):498-504. doi: 10.1007/s002800051124. PMID 10550571
- [Result] Bernstein ML, Devidas M, Lafreniere D, Souid AK, Meyers PA, Gebhardt M, Stine K, Nicholas R, Perlman EJ, Dubowy R, Wainer IW, Dickman PS, Link MP, Goorin A, Grier HE; Pediatric Oncology Group; Children's Cancer Group Phase II Study 9457; Children's Oncology Group. Intensive therapy with growth factor support for patients with Ewing tumor metastatic at diagnosis: Pediatric Oncology Group/Children's Cancer Group Phase II Study 9457--a report from the Children's Oncology Group. J Clin Oncol. 2006 Jan 1;24(1):152-9. doi: 10.1200/JCO.2005.02.1717. PMID 16382125
- [Result] Souid AK, Newton GL, Dubowy RL, Fahey RC, Bernstein ML. Determination of the cytoprotective agent WR-2721 (Amifostine, Ethyol) and its metabolites in human blood using monobromobimane fluorescent labeling and high-performance liquid chromatography. Cancer Chemother Pharmacol. 1998;42(5):400-6. doi: 10.1007/s002800050836. PMID 9771955